CLINICAL TRIAL: NCT03237091
Title: Enhancing Corticospinal Excitability to Improve Functional Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 723
Record Dates: First submitted 2017-07-24; First posted 2017-08-02 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Spinal Cord Injuries; Tetraplegia
Keywords: non-invasive brain stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Intervention Model Description: This is a a randomized, sham-controlled crossover study in which all participants will participate in a single session of each type of intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- bihemispheric transcranial pulsed current stimulation (tPCS) (Experimental)
  Interventions: Other: bihemispheric transcranial pulsed current stimulation (tPCS)
- unihemispheric transcranial pulsed current stimulation (tPCS) (Experimental)
  Interventions: Other: unihemispheric transcranial pulsed current stimulation (tPCS)
- bihemispheric transcranial direct current stimulation (tDCS) (Experimental)
  Interventions: Other: bihemispheric transcranial direct current stimulation (tDCS)
- unihemispheric transcranial direct current stimulation (tDCS) (Experimental)
  Interventions: Other: unihemispheric transcranial direct current stimulation (tDCS)
- sham-control (Active Comparator)
  Interventions: Other: sham-control

INTERVENTIONS:
Other: bihemispheric transcranial pulsed current stimulation (tPCS) — Two sets of sponge electrodes (one set placed on each side of the head) will be placed on the participant's head. The transcranial electrical stimulator will apply unidirectional, positive pulses of current separated by brief interpulse intervals to the scalp via the sponges for 30 minutes.
  Arms: bihemispheric transcranial pulsed current stimulation (tPCS)
Other: unihemispheric transcranial pulsed current stimulation (tPCS) — One set of sponge electrodes will be placed on the participant's head. The transcranial electrical stimulator will apply unidirectional, positive pulses of current separated by brief interpulse intervals to the scalp via the sponges for 30 minutes.
  Arms: unihemispheric transcranial pulsed current stimulation (tPCS)
Other: bihemispheric transcranial direct current stimulation (tDCS) — Two sets of sponge electrodes (one set placed on each side of the head) will be placed on the participant's head. The transcranial electrical stimulator will apply continuous, direct current to the scalp via the sponges for 30 minutes.
  Arms: bihemispheric transcranial direct current stimulation (tDCS)
Other: unihemispheric transcranial direct current stimulation (tDCS) — One set of sponge electrodes will be placed on the participant's head. The transcranial electrical stimulator will apply continuous, direct current to the scalp via the sponges for 30 minutes.
  Arms: unihemispheric transcranial direct current stimulation (tDCS)
Other: sham-control — Sponge electrodes will be placed on the participant's head. The transcranial electrical stimulator will apply stimulation to the scalp via the sponges for 1-2 minutes. The stimulator will then be turned off.
  Arms: sham-control

SUMMARY:
Research indicates that increasing brain excitability might help improve hand function in people with spinal cord injury. Brain stimulation that uses electrodes placed on the surface of the scalp (also called "non-invasive brain stimulation") increases brain excitability and has the potential to make it easier for the brain and nervous system to respond to arm and hand training. The purpose of this study is to compare four different types of stimulation for increasing brain excitability to determine which types are best for helping people with tetraplegia improve their ability to use their arms and hands. To fully evaluate the value of brain stimulation on arm and hand function, the investigators will also evaluate the effect of sham (fake) stimulation. Each participant will receive a single session of each of the five types of stimulation being tested.

DETAILED DESCRIPTION:
Restoration of upper extremity function is often the top rehabilitation goal for persons who have sustained a cervical spinal cord injury (SCI). Following SCI, beyond the disruption caused by the injury itself, maladaptive cortical reorganization further limits descending corticospinal drive. Therefore, therapies aimed at increasing the descending drive provided by corticospinal and other descending supraspinal tracts could be beneficial adjuncts to commonly used rehabilitation therapies. While many rehabilitation research strategies for improving function following SCI target the spinal circuitry, relatively few rehabilitative approaches are directed toward promoting supraspinal neuroplasticity to reduce impairment by increasing volitional control. Spectacular high-tech interventions and elegant high-tech outcome measures generate a great deal of excitement in the scientific world. However, the technological investment and training required for these approaches and the questionable clinical meaningfulness of the outcomes is a major limitation to their real-world value.

Transcranial direct current stimulation (tDCS) is a clinically accessible form of non-invasive brain stimulation (NIBS) that has been shown to improve upper extremity function in persons with SCI. Clinical accessibility and the potential for prolonged modulation of cortical excitability make tDCS is an attractive tool for non-invasive modulation of corticospinal excitability.

Beyond traditional tDCS, intriguing recent studies in non-disabled individuals suggest a novel form of NIBS, transcranial pulsed current stimulation (tPCS), may be more effective for inducing changes in corticospinal excitability. tPCS utilizes unidirectional, positive pulses of current separated by brief interpulse intervals rather than continuous direct current. Some evidence from our lab and others indicates that patterned stimulation has a larger influence on neural excitability than uniform stimulation.

Importantly, the efficacy of NIBS is dependent upon stimulation site. Since persons with tetraplegia have bimanual impairments, it has been suggested that bihemispheric anodal (excitatory) tDCS may be of value. Bihemispheric anodal tDCS has been studied in non-disabled individuals; this approach was found to be safe and was associated with improved bimanual control. However, the value of this approach has not previously been assessed in persons with tetraplegia.

The investigators propose a randomized, sham-controlled crossover study in which two forms of NIBS (tDCS and tPCS) will be compared with a sham-control intervention to determine their relative efficacy for improving upper extremity strength and motor control (Aim 1) and corticospinal excitability (Aim 2) in individuals with chronic (≥ 6 months) tetraplegia. The efficacy of two different stimulation montages, uni- and bihemispheric, will also be compared (Aim 3). Subjects will receive a single session of each NIBS condition (unihemispheric tDCS, bihemispheric tDCS, unihemispheric tPCS, bihemispheric tPCS) and a sham-control condition.

ELIGIBILITY:
Inclusion Criteria:

* Cervical (neurological level C1-C8) SCI occurring more than 6 months ago
* Any severity classification (ASIA/ISNCSCI A, B, C, D)
* Self-reported functional limitation in at least one upper limb
* Ability to voluntarily move thumb or index finger (visible twitch) of both upper limbs
* Ability and willingness to consent to participate in the study and authorize use of protected health information

Exclusion Criteria:

* Pacemaker or metal implant in the head
* History of seizure
* History of frequent or severe headaches
* Damage to the nerves of the arms/hands (lower motor neuron damage) as documented in medical record, per participant report, or during in-person screening
* Prior tendon or nerve transfer surgery
* Severe pain or hypersensitivity of the arm/hand that would limit participation in arm and hand training
* Severe contractures of the arm/hand that would limit participation in arm and hand training
* Current pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Motor Control & Strength | Through study completion, up to 5 weeks
  The motor control outcome measure evaluates how quickly the participant can move their fingers. Participants will tap their thumb or index finger as fast as possible for 10 seconds at a time while a sensor counts the number of taps. The strength outcome measure evaluates the participant's hand strength. Participants will use their thumb and index finger to pinch a hand-held device that measures their strength.
Change from Baseline Corticospinal Excitability | Through study completion, up to 5 weeks
  This outcome measure evaluates communication between the participant's brain and spinal cord. The skin over the muscles of both arms and hands will be cleaned with an alcohol swab and a mildly abrasive paste (similar to the feel of toothpaste). Sensors that detect muscle activity will be placed over these sites. Pulses of stimulation will be applied to the participant's head using a type of non-invasive brain stimulation called transcranial magnetic stimulation (TMS). This stimulation will activate the brain regions that control arm and hand movement. The strength of the stimulation will be increased until it causes the muscles of the arm and hand to twitch, and the size of the muscle response will be recorded with the sensors placed over the muscles.

SECONDARY OUTCOMES:
Stimulation Questionnaire | Through study completion, up to 5 weeks
  This outcome measure evaluates the participant's perception of stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States